CLINICAL TRIAL: NCT06497491
Title: A Single-blind Randomized Study of the Efficacy and Safety of the GNR-086 (Canakinumab Proposed Biosimilar) in Comparison With the Ilaris®, Conducted in Parallel Groups of Patients With Adult-onset Still's Disease
Brief Title: An Efficacy and Safety Study of GNR-086 (Canakinumab Biosimilar) and Ilaris® in Patients With Adult-onset Still's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AO GENERIUM (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CAN-AOSD-III
Record Dates: First submitted 2024-07-05; First posted 2024-07-11 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Still's Disease Adult Onset
Keywords: canakinumab; humanized monoclonal antibodies; safety; Still's disease adult onset; equivalence; biosimilar; American College of Rheumatology (ACR); DAS28; disease-modifying anti-rheumatic drugs (DMARDs); European League Against Rheumatism (EULAR); immunogenicity
MeSH Terms: conditions — Wissler's Syndrome | interventions — canakinumab

STUDY DESIGN:
Who Masked: Participant
Masking Description: Analitial laboratory to assess imunogenicity
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- GNR-086 (Experimental): canakinumab biosimilar
  Interventions: Biological: GNR-086
- Ilaris® (Active Comparator): canakinumab
  Interventions: Biological: Ilaris®

INTERVENTIONS:
Biological: GNR-086 — GNR-086 is administered as a subcutaneous injection at a dose of 4 mg/kg once every 4 weeks for 24 weeks.
  Other Names: canakinumab biosimilar
  Arms: GNR-086
Biological: Ilaris® — Ilaris® is administered as a subcutaneous injection at a dose of 4 mg/kg once every 4 weeks for 24 weeks.
  Other Names: canakinumab
  Arms: Ilaris®

SUMMARY:
This is a randomized single-blind comparative parallel group study of the efficacy and safety of canakinumab biosimilar GNR-086 (JSC "GENERIUM", Russia) and Ilaris® (Novartis Pharma Stein AG, Switzerland) in the treatment of patients with adult-onset Still's disease. Participants will receive a subcutaneous canakinumab 4 mg/kg every 4 weeks. The treatment duration is 24 weeks following with the study extension.

DETAILED DESCRIPTION:
GNR-086 is being developed as a proposed biosimilar to Ilaris®, a lyophilisate for the preparation of a solution for subcutaneous administration.

Canakinumab is a fully human monoclonal antibody of the immuniglobulin G1 (IgG1(kappa)) isotype that binds specifically and with high affinity to interleukin-1β (IL-1β). Canakinumab, by binding to human IL-1β, blocks the interaction of this cytokine with its receptors, thereby functionally neutralizing the biological activity of this cytokine, without preventing either the binding of the natural inhibitor IL-1Ra, or the binding of IL-1α to IL-1 receptors. IL-1β is recognized as one of the main pro-inflammatory cytokines in various inflammatory conditions.

This III phase study is aimed to compare the efficacy, safety and immunogenicity of GNR-086 and Ilaris®. The study will enroll patients with the confirmed diagnosis of adult-onset Still's disease in accordance with the classification criteria of Yamaguchi M. et al. (J. Rheumatology, 1992), and the duration of the disease at least 2 months before inclusion into the study. 148 paitnts will be randomised 2:1 to receive either GNR-098 or Ilaris®. Participants will receive canakinumab 4 mg/kg suncutaneously every 4 weeks for 24 weeks following the study extension.

ELIGIBILITY:
Inclusion Criteria:

* Availability of written informed consent obtained from the patient before the start of any procedures related to the study.
* Male and female patients aged 18-75 years, inclusive, at the time of signing the informed consent form.
* Patients with a documented diagnosis of adult Still's disease in accordance with the classification criteria of Yamaguchi M. et al. (J. Rheumatology, 1992) and the duration of the disease is at least 2 months before signing the Informed Consent Form.
* Disease activity ≥2.6 according to DAS28-ESR.
* No change in the dosing regimen of methotrexate (maximum 20 mg/m2/week) or other immunosuppressive agent for at least 6 weeks before randomization and/or no change in the dosing regimen of one nonsteroidal anti-inflammatory drug (NSAID) as treatment for adult Still's disease for at least 14 days before randomization and/or no change in the dosage regimen of the glucocorticosteroid drug for at least 7 days before randomization.
* Negative result of intradermal test with tuberculosis allergen / IGRA test at screening or within 6 months before screening. Patients with missing screening data can only be included in the study if they undergo immunodiagnosis of tuberculosis infection and the result is negative.
* Agreement to adhere to adequate methods of contraception throughout the study and for 3 months after the end of canakinumab therapy.

Exclusion Criteria:

* Diagnosis of macrophage activation syndrome (MAS) within the last 3 months.
* History of hypersensitivity to the active substance or other components of the study or reference drug.
* Acute infectious diseases within 14 days before randomization.
* Immunization with any live vaccine within 3 months before randomization.
* Concomitant diseases and conditions that, in the opinion of the Investigator and/or Sponsor, jeopardize the safety of the patient during participation in the study, or which will influence the analysis of safety data.
* Blood donation or blood loss (450 ml of blood or more) less than 2 months before the start of the study.
* Pregnancy or breastfeeding.
* History of tuberculosis (except for successfully treated primary tuberculosis complex no later than 6 months before randomization).
* Use of the following treatments before randomization: anakinra within 1 week before randomization; etanercept within 6 weeks before randomization; tocilizumab within 8 weeks before randomization; sarilumab within 6 weeks before randomization; olokizumab for 8 weeks before randomization; adalimumab within 10 weeks before randomization; golimumab within 16 weeks before randomization; rituximab within 26 weeks before randomization; leflunomide within 6 weeks before randomization; cyclosporine within 4 weeks before randomization; intravenous immunoglobulin within 8 weeks before randomization; growth hormone within 4 weeks before randomization; intra-articular, periarticular, intravenous, intramuscular administration of glucocorticosteroids within 4 weeks before randomization; any other unapproved drugs within 5 half-lives before randomization.
* Drug dependence on drugs and potent drugs and/or alcohol dependence.
* Positive test results for hepatitis B or C, HIV or syphilis.
* Unwillingness or inability to comply with the recommendations prescribed by this protocol.
* Identification during screening of other diseases/conditions not listed above that, in the opinion of the physician-researcher, prevent the inclusion of the patient in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2023-12-12 (Actual); Primary Completion 2025-05-29 (Actual); Study Completion 2025-07-10 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with a clinically significant (>1.2 points) decrease in the Disease Activity Score-28 for Rheumatoid Arthritis with Erythrocyte Sedimentation Rate (DAS28-ESR) | Week 12
  A composite index and takes into account the following items: Tender joint count (number of tender joints; 0-28); swollen joint count (number of swollen joints; 0-28); ESR (mm/h) and Global Health (Patient's Global Assessment of Disease Activity; from 0=best to 100=worst). Thus, given the reliability, validity, and ability of DAS28 to discriminate the severity of joint involvement, this index has been used in other rheumatic diseases characterized by rheumatoid artritis (RA)-like poly-articular involvement. Of note, a DAS28 score > 5.1 implies active disease, ≤3.2 low disease activity, and <2.6 remission. Moderate/high disease activity is defined as a DAS28 higher than 3.2.

SECONDARY OUTCOMES:
Change in DAS28-ESR/C-reactive protein (CRP) score | Week 24
  A composite index and takes into account the following items: Tender joint count (number of tender joints; 0-28); swollen joint count (number of swollen joints; 0-28); ESR (mm/h) / CRP (mg/l) and Global Health (Patient's Global Assessment of Disease Activity; from 0=best to 100=worst). Thus, given the reliability, validity, and ability of DAS28 to discriminate the severity of joint involvement, this index has been used in other rheumatic diseases characterized by RA-like poly-articular involvement.
Proportion of patients with an American College of Rheumatology score (ACR) 30/50/70/90/100 response without fever associated with the underlying disease during the 7 days preceding the day of assessment | Week 24
  The ACR30/50/70/90/100 response: greater than or equal to (>/=) 30/50/70/90/100 percent (%) improvement in TJC and SJC (28 assessed joints), and 30/50/70/90/100 % improvement in 3 of the following 5 criteria, respectively: 1) physician's assessment Global Disease Activity (PhGDA), 2) Patients assessment Global Disease Activity (PtGDA), 3) participant's assessment of pain, 4) participant's assessment of functional disability via a health assessment questionnaire, and 5) CRP or ESR
Area under the curve (AUC) of the disease activity rate (ACR) | Week 24
  ACR response criteria measure percentage reduction in 68 painful joints, percentage reduction in 66 swollen joints, and percentage improvement in at least three of the following: Patients assessment Global Disease Activity (PtGDA), physician's assessment Global Disease Activity (PhGDA), Patient Pain Assessment , assessment according to the health assessment questionnaire disability index (HAQ-DI), CRP concentration value.
Proportion of Participants With European League Against Rheumatism (EULAR) Response Based on DAS28 | Week 24
  The DAS28-based EULAR response criteria were used to measure individual response as none, good, and moderate, depending on the extent of change from baseline and the level of disease activity reached. Good responders: change from baseline >1.2 with DAS28 </=3.2; moderate responders: change from baseline >1.2 with DAS28 >3.2 to </=5.1 or change from baseline >0.6 to </=1.2 with DAS28 </=5.1; non-responders: change from baseline </=0.6 or change from baseline >0.6 and </=1.2 with DAS28 >5.1
Area under the curve (AUC) of CRP concentration | Week 24
  CRP values standardized to a normal range
Area under the curve (AUC) of ESR | Week 24
  ESR values standardized to a normal range
Area under the curve (AUC) of ferritin levels | Week 24
  Ferritin values standardized to a normal range
Proportion of patients with no rash within 24 hours before the end of the 1st week of treatment; and within 7 days before all subsequent visits | Week 24
  The absence or presence of skin rash assessed based on physical exam findings including whether it is typical or atypical
Proportion of patients with fever associated with the underlying disease during 24 weeks of treatment | Week 24
  Absence of fever associated with the underlying disease during the 7 days preceding the visit day visit was assessed. Fever is defined as an increase in body temperature ≥38.0 °C
Proportion of patients who had exacerbations | Week 24
  Increasing disease activity is defined as the appearance of signs of systemic activity, defined as any of the "major" Yamaguchi M. classification criteria (fever >39°C intermittent for ≥1 week; arthralgias ≥2 weeks; characteristic rash; white blood cells >10,000 in mm3 (>80% granulocytes)), as well as an increase in CRP and/or ferritin levels ≥ 3 times normal.

CONTACTS AND LOCATIONS:
Overall Officials: Oksana A. Markova, MD, Study Chair — JSC GENERIUM
Locations (17):
- Russia (17):
  - State budgetary healthcare institution "Chelyabinsk Regional Clinical Hospital", Chelyabinsk, Chelyabinsk Oblast
  - Limited Liability Company "Medical Center "Revma-Med", Kemerovo, Kemerovo Oblast
  - Limited Liability Company "OLLA-MED", Moscow, Moscow
  - Federal State Budgetary Institution "Research Institute of Rheumatology named after V.A. Nasonova", Moscow, Moscow
  - State budgetary healthcare institution of the city of Moscow "City Clinical Hospital No. 52 of the Moscow Health Department" (GBUZ "City Clinical Hospital No. 52 DZM"), Moscow, Moscow
  - Federal State Autonomous Educational Institution of Russian National Research Medical University named after. N. I. Pirogova, Moscow, Moscow
  - Federal State Autonomous Educational Institution of Russian National Research Medical University named after. N.I. Pirogov Ministry of Health of Russia Separate structural unit "Russian Gerontological Scientific and Clinical Center", Moscow, Moscow
  - Limited Liability Company "Medical Center "Healthy Family", Novosibirsk, Novosibirsk Oblast
  - Federal State Budgetary Educational Institution of Higher Education Orenburg State Medical University of the Ministry of Health of Russia, Orenburg, Orenburg Oblast
  - Limited Liability Company "Medical Technologies" LLC "Medical Technologies", Saint Petersburg, Sankt-Peterburg
  - Limited Liability Company "Ex Seven Clinical Research", Saint Petersburg, Sankt-Peterburg
  - Limited Liability Company "Interleukin", Saint Petersburg, Sankt-Peterburg
  - State Budgetary Healthcare Institution Leningrad area Clinical Hospital, Saint Petersburg, Sankt-Peterburg
  - Private foundation "RZD-Medicine" Smolensk", Smolensk, Smolensk Oblast
  - Limited Liability Company "BioMed", Vladimir, Vladimirskaya Oblast’
  - State health care institution city clinical hospital №25, Volgograd, Volgograd Oblast
  - State Budgetary Healthcare Institution "Clinical Hospital No. 2", Yaroslavl, Yaroslavl Oblast

IPD SHARING:
Plan to Share IPD: No